CLINICAL TRIAL: NCT04121221
Title: A Phase III Study in Subjects With Relapsing Forms of Multiple Sclerosis (RMS) to Asses Efficacy, Safety and Tolerability of GA Depot, a Long Acting IM Injection of Glatiramer Acetate, Once Monthly Compared to Placebo
Brief Title: A Study to Asses Efficacy, Safety and Tolerability of Monthly Long-acting IM Injection of GA Depot in Subjects With RMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mapi Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mapi GA Depot Phase III - 001
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; RMS; GA Depot; Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: During the placebo controlled period subjects will receive either 40mg of GA Depot or matching placebo, IM, once every 4 weeks, for a total of 13 times.
  Subjects who complete the PC period of the study will be offered to continue into the open label period for an additional 52 weeks, in which all subjects will receive 40mg of GA Depot IM once every 4 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GA Depot (Experimental): Monthly IM injection
  Interventions: Drug: GA Depot
- Placebo (Placebo Comparator): Monthly IM injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GA Depot — Long acting intramuscular injection of glatiramer acetate, once every 4 weeks
  Arms: GA Depot
Other: Placebo — IM injection once every 4 weeks
  Arms: Placebo

SUMMARY:
A multinational, multicenter, randomized, Phase III, double blind, parallel group, placebo controlled study in subjects with Relapsing Forms of Multiple Sclerosis (RMS) to assess the efficacy, safety and tolerability of GA Depot, a long acting IM injection of glatiramer acetate, administered once every four weeks

DETAILED DESCRIPTION:
A total of 1000 subjects are planned to be randomized into this study to receive treatment with GA Depot or with matching placebo.

During the placebo controlled period (PC period, the first 52 weeks of the study immediately after randomization) subjects will receive either 40mg of GA Depot or matching placebo, IM, once every 4 weeks, for a total of 13 times.

Subjects who complete the PC period of the study will be offered to continue into the open label period (OL period) for an additional 52 weeks, in which all subjects will receive 40mg of GA Depot IM once every 4 weeks.

ELIGIBILITY:
Inclusion criteria:

1. Adult subjects between 18-55 years of age, inclusive.
2. Subjects able to provide signed written informed consent.
3. Subjects must be willing and able to comply with the protocol requirements for the duration of the study.
4. MS diagnosis fulfilling the 2017 McDonald Criteria.
5. Subjects should be ambulatory with an EDSS score of 0-5.5 at screening and baseline visits. EDSS score will be determined by a separate, blinded trained EDSS rater.
6. Subjects should be relapse free and neurologically stable from one month before screening visit and from screening visit to baseline visit.
7. No systemic corticosteroid treatment or ACTH within one month prior to screening visit.
8. Subjects must have experienced at least one of the following:

   i. At least one documented relapse in the 12 months prior to screening. ii. At least two documented relapses in the 24 months prior to screening. iii. One documented relapse between 12 and 24 months prior to screening, with at least one documented T1-Gd enhancing lesion in MRI performed within 0-12 months before screening.
9. Women capable of child bearing must have a negative urine pregnancy test at screening and baseline visit and use an adequate contraceptive method throughout the study.

Exclusion criteria:

1. Use of experimental / investigational drug, and / or participation in drug clinical studies within the 6 months prior to screening.
2. Any off-label drug use for MS treatment such as high dose simvastatin and biotin within 6 months prior to screening.
3. Previous use of immunosuppressant including Mitoxantrone, Alemtuzumab, Cladribine or any other cytotoxic agent within 5 years.
4. Previous use of Natalizumab or any anti-B cell agent within 9 months prior to screening.
5. Previous use of Fingolimod or any other sphingosine-1-phosphate receptor modulator, Dimethyl Fumarate, Diroximel Fumarate (DRF), or Monomethyl fumarate within 2 months prior to screening. Subjects will be excluded if they do not have a lymphocyte count of above 1,000/mm3 at screening.
6. Previous use of Teriflunomide within 12 months if no accelerated elimination procedure was used.
7. Previous treatment with immunomodulators (including IFNβ 1a and 1b, and IV Immunoglobulin (IVIg) within 2 months prior to screening.
8. Previous use of GA or any other glatiramoid.
9. Chronic (more than 30 consecutive days) systemic (IV, PO or IM) corticosteroid treatment within 6 months prior to screening visit.
10. Previous total body irradiation or total lymphoid irradiation.
11. Previous stem-cell treatment, autologous bone marrow transplantation or allogeneic bone marrow transplantation.
12. Subjects with a clinically significant or unstable medical, psychiatric, or surgical conditions that would preclude safe and complete study participation, as determined by medical history, physical exams, ECG and/or abnormal laboratory tests; and or subjects with an increased risk of serious Covid-19 related morbidity. Such conditions may include hepatic, renal or metabolic diseases, systemic disease, acute infection, current malignancy, or recent history (5 years) of malignancy, major psychiatric disorder, history of drug and/or alcohol abuse and allergies that could be detrimental according to the investigator's judgment.
13. Subjects who have >10 T1-Gd enhancing lesions at screening.
14. A known history of sensitivity to Gadolinium.
15. Inability to successfully undergo MRI scanning.
16. Pregnant or breast-feeding women.
17. Abnormal renal function.
18. Abnormal liver function.
19. History of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study article (e.g., GA, Polyglactin, PVA).
20. Positive testing or a history of positive testing for syphilis, HIV, hepatitis, or tuberculosis.
21. Known or suspected history of drug or alcohol abuse.
22. Subjects diagnosed with any systemic autoimmune disease (other than MS) that may impact the CNS with MS like lesions such as Sarcoidosis, Sjögren's syndrome, Systemic Lupus Erythematosus (SLE), Lyme disease, Antiphospholipid antibodies (APLA) syndrome, etc. Subjects with stable local/organ autoimmune disease such as psoriasis, cutaneous lupus erythematosus, thyroiditis (Hashimoto's, Grave's) etc. may be considered eligible upon the investigator's discretion.
23. Any CNS disorder other than MS that may jeopardize the subject's participation in the study.
24. Subjects with uncontrolled diabetes.
25. Subjects with clotting disorders or receiving treatment with anticoagulants.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1016 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Annualized Relapse Rate (ARR) | 52 weeks
  Annualized Relapse Rate (ARR) will be derived from the total number of confirmed relapses.

SECONDARY OUTCOMES:
Changes in brain MRI (number of T1 lesions) | 52 weeks
  Cumulative number of new enhancing lesions on T1-weighted images as compared to baseline.
Changes in brain MRI (number of T2 lesions) | 52 weeks
  Cumulative number of new or newly enlarging hyperintense T2 lesions as compared to baseline.
Hyperintense T2-lesion volume change | 52 weeks
  Change from baseline to Week 52 in hyperintense T2-lesion volume.
Enhancing T1-lesion volume change | 52 weeks
  Change from baseline to Week 52 in enhancing T1-lesion volume.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Popper, MD, Study Director — Mapi Pharma Ltd.; Aaron E. Miller, Prof. MD, Principal Investigator — Mount Sinai School of Medicine, New York, US
Locations (112):
- United States (11):
  - Mapi Pharma Research site 08, Birmingham, Alabama
  - Mapi Pharma Research site 11, Cullman, Alabama
  - Mapi Pharma Research site 15, Pasadena, California
  - Mapi Pharma Research site 14, Denver, Colorado
  - Mapi Pharma Research site 12, Washington D.C., District of Columbia
  - Mapi Pharma Research site 17, Homestead, Florida
  - Mapi Pharma Research site 09, Miami, Florida
  - Mapi Pharma Research site 01, Northbrook, Illinois
  - Mapi Pharma Research site 02, Detroit, Michigan
  - Mapi Pharma Research site 13, Westerville, Ohio
  - Mapi Pharma Research site 04, Round Rock, Texas
- Belarus (6):
  - Mapi Pharma Research site 02, Homyel
  - Mapi Pharma Research site 04, Minsk
  - Mapi Pharma Research site 05, Minsk
  - Mapi Pharma Research site 06, Minsk
  - Mapi Pharma Research site 01, Vitebsk
  - Mapi Pharma Research site 07, Vitebsk
- Bosnia and Herzegovina (4):
  - Mapi Pharma Research site 04, Banja Luka
  - Mapi Pharma Research site 06, Bihać
  - Mapi Pharma Research site 01, Sarajevo
  - Mapi Pharma Research site 03, Tuzla
- Bulgaria (19):
  - Mapi Pharma Research site 14, Haskovo
  - Mapi Pharma Research site 10, Pazardzhik
  - Mapi Pharma Research site 01, Pleven
  - Mapi Pharma Research site 02, Pleven
  - Mapi Pharma Research site 03, Pleven
  - Mapi Pharma Research site 07, Pleven
  - Mapi Pharma Research site 12, Plovdiv
  - Mapi Pharma Research site 18, Rousse
  - Mapi Pharma Research site 04, Sofia
  - Mapi Pharma Research site 05, Sofia
  - Mapi Pharma Research site 06, Sofia
  - Mapi Pharma Research site 08, Sofia
  - Mapi Pharma Research site 11, Sofia
  - Mapi Pharma Research site 13, Sofia
  - Mapi Pharma Research site 15, Sofia
  - Mapi Pharma Research site 16, Sofia
  - Mapi Pharma Research site 19, Sofia
  - Mapi Pharma Research site 09, Veliko Tarnovo
  - Mapi Pharma Research site 17, Vratsa
- Mapi Pharma Research site 01, Tallinn, Estonia
- Georgia (9):
  - Mapi Pharma Research site 01, Tbilisi
  - Mapi Pharma Research site 02, Tbilisi
  - Mapi Pharma Research site 03, Tbilisi
  - Mapi Pharma Research site 04, Tbilisi
  - Mapi Pharma Research site 05, Tbilisi
  - Mapi Pharma Research site 06, Tbilisi
  - Mapi Pharma Research site 07, Tbilisi
  - Mapi Pharma Research site 08, Tbilisi
  - Mapi Pharma Research site 09, Tbilisi
- Israel (2):
  - Mapi Pharma Research site 01, Safed
  - Mapi Pharma Research site 02, Tel Aviv
- Moldova (2):
  - Mapi Pharma Research site 01, Chisinau
  - Mapi Pharma Research site 02, Chisinau
- Russia (28):
  - Mapi Pharma Research site 29, Barnaul
  - Mapi Pharma Research site 27, Bryansk
  - Mapi Pharma Research site 23, Chelyabinsk
  - Mapi Pharma Research site 01, Kazan'
  - Mapi Pharma Research site 19, Kemerovo
  - Mapi Pharma Research site 24, Krasnodar
  - Mapi Pharma Research site 03, Moscow
  - Mapi Pharma Research site 13, Moscow
  - Mapi Pharma Research site 14, Moscow
  - Mapi Pharma Research site 21, Moscow
  - Mapi Pharma Research site 25, Moscow
  - Mapi Pharma Research site 28, Moscow
  - Mapi Pharma Research site 02, Nizhny Novgorod
  - Mapi Pharma Research site 07, Nizhny Novgorod
  - Mapi Pharma Research site 10, Nizhny Novgorod
  - Mapi Pharma Research site 11, Novosibirsk
  - Mapi Pharma Research site 06, Perm
  - Mapi Pharma Research site 22, Pyatigorsk
  - Mapi Pharma Research site 08, Rostov-on-Don
  - Mapi Pharma Research site 09, Saint Petersburg
  - Mapi Pharma Research site 18, Saint Petersburg
  - Mapi Pharma Research site 20, Saint Petersburg
  - Mapi Pharma Research site 05, Samara
  - Mapi Pharma Research site 26, Saransk
  - Mapi Pharma Research site 15, Smolensk
  - Mapi Pharma Research site 16, Tyumen
  - Mapi Pharma Research site 04, Ufa
  - Mapi Pharma Research site 17, Ulyanovsk
- Ukraine (30):
  - Mapi Pharma Research site 32, Cherkasy
  - Mapi Pharma Research site 06, Chernihiv
  - Mapi Pharma Research site 11, Chernivtsi
  - Mapi Pharma Research site 03, Dnipro
  - Mapi Pharma Research site 04, Dnipro
  - Mapi Pharma Research site 24, Dnipro
  - Mapi Pharma Research site 18, Ivano-Frankivsk
  - Mapi Pharma Research site 26, Ivano-Frankivsk
  - Mapi Pharma Research site 27, Ivano-Frankivsk
  - Mapi Pharma Research site 09, Kharkiv
  - Mapi Pharma Research site 10, Kharkiv
  - Mapi Pharma Research site 08, Kherson
  - Mapi Pharma Research site 21, Kyiv
  - Mapi Pharma Research site 25, Kyiv
  - Mapi Pharma Research site 28, Kyiv
  - Mapi Pharma Research site 29, Kyiv
  - Mapi Pharma Research site 17, Lutsk
  - Mapi Pharma Research site 12, Lviv
  - Mapi Pharma Research site 13, Lviv
  - Mapi Pharma Research site 23, Lviv
  - Mapi Pharma Research site 05, Odesa
  - Mapi Pharma Research site 14, Poltava
  - Mapi Pharma Research site 34, Ternopil
  - Mapi Pharma Research site 31, Uzhhorod
  - Mapi Pharma Research site 16, Vinnitsa
  - Mapi Pharma Research site 01, Zaporizhzhya
  - Mapi Pharma Research site 02, Zaporizhzhya
  - Mapi Pharma Research site 07, Zaporizhzhya
  - Mapi Pharma Research site 20, Zaporizhzhya
  - Mapi Pharma Research site 33, Zhytomyr